CLINICAL TRIAL: NCT07265778
Title: Multicenter, Randomized, Subject & Independent Evaluator-blind, Split-face, Medical Device Pivotal Study to Evaluate the Efficacy and Safety of Injection With JTM102 as Compared to Juvederm VOLUMA With Lidocaine for Temporary Restoring the Mid-face Volume
Brief Title: Clinical Investigation for Evaluating the Safety and Efficacy of JTM102 to Mid Face Volume Deficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jetema Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JT-D-102-01
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Mid Face Volume Deficit
Keywords: mid-face volume; HA filler

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JTM102 (Experimental): HA filler with lidocaine
  Interventions: Device: JTM102
- Juverderm Voluma with Lidocaine (Active Comparator): HA filler with lidocaine
  Interventions: Device: Juvederm VOLUMA with Lidocaine

INTERVENTIONS:
Device: JTM102 — Sodium Hyaluronate 20mg/ml Lidocaine Hydrochloride 03.%
  Arms: JTM102
Device: Juvederm VOLUMA with Lidocaine — Sodium Hyaluronate 20mg/ml Lidocaine Hydrochloride 0.3%
  Arms: Juverderm Voluma with Lidocaine

SUMMARY:
This study is clinical investigation for evaluating safety and efficacy of JTM102 on temporary correction of mid-face volume deficiency

DETAILED DESCRIPTION:
This study is Multicenter, Randomized, Subject & Independent Evaluator-blind, Split-face, Medical Device Pivotal study to evaluate the efficacy and safety of injection with JTM102 as compared to Juvederm VOLUMA with Lidocaine for temporary restoring the mid-face volume

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily agree to participate in this clinical trial.
* Adults aged 19 to 65 years.
* Subjects who desire temporary improvement of mid-face volume and whose Mid-face Volume Deficit Scale (MFVDS, 5-point scale) score for the mid-face volume restoration meets eligibility criteria
* Subjects who agree to discontinue all dermatological treatments or procedures for the face during the clinical trial period, including wrinkle improvement treatments such as fillers, botulinum toxin, laser therapy, chemical peels, and cosmetic surgeries, except for the investigational medical device application.
* Subjects who use medically acceptable contraception methods throughout the clinical trial period (pregnant or breastfeeding women are excluded).
* Subjects who understand and can comply with the study instructions and can participate for the entire duration of the clinical trial.

Exclusion Criteria:

* History or concurrent conditions included in exclusion criteria
* History of procedures (including surgery) included in exclusion criteria
* Use of medications that may affect evaluation of the investigational device:
* Any other conditions judged by the investigator as inappropriate for participation in this clinical trial.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MFVDS | 24 weeks after final application of the investigational medical device
  Improvement rate in the Mid-Face Volume Deficit Scale (MFVDS), as assessed by independent photographic evaluators, compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chungang University Hospital, Seoul, South Korea